CLINICAL TRIAL: NCT04567641
Title: Impact of Early Enteral & Parenteral Nutrition on Post-operative Outcome After Abdominal Surgery
Brief Title: Early Nutrition Impact on Post Abdominal Surgery Outcome
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Farouk, clinical professor, Cairo University
Other Study IDs: MS-311-2016
Record Dates: First submitted 2020-09-20; First posted 2020-09-28 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Postoperative Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Enteral Nutrition
  Interventions: Dietary Supplement: postoperative nutrition
- Parenteral nutrition
  Interventions: Dietary Supplement: postoperative nutrition

INTERVENTIONS:
Dietary Supplement: postoperative nutrition — Forty patients (50%) received enteral nutrition 6 hours after surgical procedures and 40 patients (50%) received parenteral nutrition 6 hours after surgical procedures.

SUMMARY:
Introduction: Nutritional support is a vital therapy of most surgical patients. Early initiation via the enteral route has a significant effect on postoperative recovery. The prognostic role of CRP and albumin can be explained by their abilities to reflect inflammation in the acute phase in critical settings and assess the nutritional status of critically ill patients, respectively. This indicates the prognostic value of the CRP/ALB ratio in postoperative patients admitted to the ICU.

Aim of work: Determine the effect of early enteral & parenteral nutrition on ICU outcome & nutritional status in postoperative abdominal surgical patients and investigate the effect of enteral & parenteral nutrition on CRP/albumin ratio as an inflammatory marker & its correlation with SOFA score.

Methods: A prospective cohort non randomized study included 80 postoperative abdominal surgical patients at Critical Care Department, Cairo University over one year duration. Forty patients (50%) received enteral nutrition 6 hours after surgical procedures and 40 patients (50%) received parenteral nutrition 6 hours after surgical procedures. Nutritional status and inflammatory markers were screened. All patients were followed up during the ICU stay & up to 3 months. SOFA scoring was done every 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* postoperative abdominal surgical patients at Critical Care Department, Cairo University over one year duration.
* age between 18-80 years

Exclusion Criteria:

* renal failure
* liver failure
* extensive burns
* hemodynamic instability.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included patients with age more than 18 years underwent major abdominal surgeries.
  Pre-operative nutrition screening was done using Nutritional risk screening (NRS 2000).
  Patients were divided into two groups: Group A: 40 patients (50%) received enteral nutrition 6 hours after surgical procedure & Group B: 40 patients (50%) received parenteral nutrition 6 hours after surgical procedure according to the surgeons preference.
  Enteral feeding in group (A) was started 6 hours postoperatively via ryle tube or feeding jejunostomy including proteins (1.5 gm/kg/day) with a caloric value (4.1 kcal/gm), fat (caloric value = 9 kcal/gm) & carbohydrates.
  Parenteral feeding in group (B) was started 6 hours postoperatively using SmofKabiven Peripheral [FRESENIUS KABI] : 1200 ml , 38 gm amino acids, 34 gm lipids, 85 gm glucose, osmolarity 850 mosmol/L with total energy approximately 800Kcal.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Gastro-intestinal tolerance: vomitting or diarrhea | 7 days
  number of participants who develop nausea, vomitting or diarrhea
Refeeding syndrome; hypokalemia and hypophosphatemia | 7 days
  number of participants who develop hypokalemia and hypophosphatemia
length of ICU stay | 7 days
  measurement of days of ICU stay
duration of mechanical ventilation. | 7 days
  measurement of days of mechanical ventilation

SECONDARY OUTCOMES:
3 months survival after discharge . | 90 days
  measurement of the rate of survival within 3 months between participants
re-admission within 30 days | 30 days
  measurement of the rate of hospital re-admission within 30 days between participants